CLINICAL TRIAL: NCT05192525
Title: The Effects of a Nurse-led MHealth Program for Symptom Self-management of Breast Cancer Patients Undergoing Chemotherapy in Shanghai: a Randomized Controlled Pilot Trial
Brief Title: The Effects of a Nurse-led MHealth Program for Symptom Self-management of Breast Cancer Patients Undergoing Chemotherapy
Acronym: mChemo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hong Kong Polytechnic University (Other)
Collaborators: Ruijin Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: HSEARS20210816002
Record Dates: First submitted 2021-12-09; First posted 2022-01-14 (Actual); Last update posted 2024-10-10 (Actual); Status verified 2021-09

CONDITIONS: Breast Cancer; Chemotherapeutic Toxicity
Keywords: nurse-led; mHealth; self-management; breast cancer; chemotherapy
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: The study will be a double-blinded, randomized, controlled trial, including one intervention group (group A) and one control group (group B). The control group will be treated with routine care only. The intervention group participants will receive one core intervention "mChemotherapy", one pre-chemotherapy consultation, and two scheduled visits. "mChemotherapy" is built on the official WeChat platform of the Ruijin Breast Health Centre and includes six components: (i) self-monitoring, (ii) alerts, (iii) reminder, (iv) consultation, (v) my prescription, (vi) knowledge base. The intervention group participants will take part in an mChemotherapy program for six weeks. The intervention nurses will deliver the intervention and contact patients through this platform.
Who Masked: Participant, Outcomes Assessor
Masking Description: The control group will be blinded to the allocation results and intervention. The experimental group will be informed the procedure of intervention. Before participants sign the consent form, the results of the group random assignments will be put in opaque envelopes handed out by a nurse, who will not be involved in the allocation and intervention, to participants during their pre-chemotherapy consultation. The data collectors will be blinded to the allocation results. The nurses and research assistants arranging the process of screening participants for eligibility will not be in charge of the group allocations and intervention. The nurses who will be responsible for the control group with routine care will not be involved in the intervention or the screening and group allocations.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- mChemotherapy group (Experimental): The intervention group participants will adopt an app "mChemotherapy" to self-manage their symptoms under nurse-led supervision for six weeks.
  Interventions: Device: mChemotherapy
- Control group (No Intervention): Participants in control group will receive routine care, with no use of mChemotherapy during six weeks. Routine care is composed of a pre-chemotherapy visit and two follow-up visits. Through the Official WeChat platform, the patients in control group will be informed about the chemotherapy regimen, and chemotherapy-related symptoms and how to deal with them, during the pre-chemotherapy visit. The control group will have two scheduled visits by telephone with the follow-up nurse. Patients will be given a phone number for consulting the follow-up nurse should they have questions related to their symptoms, or concerns related to the chemotherapy. Patients in the control group cannot access the "mChemotherapy" until they have completed the pilot study.

INTERVENTIONS:
Device: mChemotherapy — The intervention is composed of one core intervention "mChemotherapy", one pre-chemotherapy consultation, and two app follow-up visits. mChemotherapy will be specifically utilized to facilitate symptom self-management for intervention group covering chemotherapy for six weeks. The mChemotherapy includes six components: (i) self-monitoring, (ii) alerts, (iii) reminder, (iv) consultation, (v) my prescription, (vi) knowledge base. Intervention group participants will be given an individual username and password to log in to the mChemotherapy platform. The intervention nurses will deliver the intervention and contact patients through this platform.
  Arms: mChemotherapy group

SUMMARY:
Breast cancer (BC) survivors will experience multiple symptoms following chemotherapy. During the pandemic of COVID-19, the closure of clinics and fear of infection lead to BC patients' challenges in self-managing their multiple symptoms in home settings. Mobile health (mHealth), without time and space limitation, plays a positive role in supporting self-management and treatment compliance. However, previous mHealth self-management studies did not report sustained beneficial effects with physician-led supervision. In oncology practice, the nurse-led model of patient self-management for breast cancer has been placed on greater emphasis. Accordingly, an innovative nurse-led supervised mHealth program was designed to support self-management for BC patients undergoing chemotherapy.

This pilot study aims to examine the feasibility and acceptability of a nurse-led mHealth-based self-management program for BC patients receiving chemotherapy, in order to provide evidence for conducting a definitive trial. The feasibility outcomes of the pilot study include subject eligibility rate, recruitment rate, and retention rate. The efficacy outcomes relate to self-efficacy (primary outcome), symptom distress and frequency, as well as health-related quality of life, and healthcare utilisation. The qualitative outcomes encompass patient- and provider-users' perceptions of the app usability and subjects' experiences of engaging in the pilot study.

DETAILED DESCRIPTION:
This nurse-led mHealth symptom self-management program is composed of one core intervention 'mChemotherapy', one pre-chemotherapy consultation, and two follow-up visits. mChemotherapy will be specifically utilized to facilitate symptom self-management for breast cancer patients covering chemotherapy.

The objectives of the pilot study are: (i) to develop an evidence-based nurse-led mHealth guideline for self-management of chemotherapy-related symptoms; (ii) to determine the usability of a nurse-led mobile application; (iii) to pilot the methodological procedures of the randomized controlled trial; (iv) to determine enrollment rate, the eligibility rate, retention rate, and dropout rate during the preliminary RCT participant recruitment and follow-up process; (v) to preliminarily test the effectiveness of this program on self-efficacy, QoL, symptom distress and symptom frequency, as well as healthcare utilization; (vi) to identify the participants' perceptions and acceptability of the pilot study; (vii) to provide suggestions and implications for a future multicentre large-scale RCT examining the definite effects of nurse-led mHealth self-management guidelines on self-efficacy, QoL, symptom distress and symptom frequency in cancer patients undergoing chemotherapy.

The pilot study aims to examine the following null hypotheses of efficacy outcomes:

The BC patients in the mHealth group will demonstrate no difference in self-efficacy, quality of life, symptom distress and symptom frequency, as well as healthcare utilization after completing the chemotherapy at week 3 and week 6 when compared to the BC patients in the control group.

ELIGIBILITY:
Inclusion Criteria:

* People who are 18 years or above
* Newly diagnosed with breast cancer
* Commencing chemotherapy and being prescribed with four cycles of a chemotherapy regimen
* Mobile phone and WeChat® users (a mobile application of Shenzhen city's Tencent computer system Co. Ltd.)
* Wi-Fi or 4G network users
* Able to read and write Chinese

Exclusion Criteria:

* People who are pregnant
* Have been diagnosed with terminal-stage breast cancer (i.e., stage IV)
* Have a history of chemotherapy
* Have been prescribed with targeted therapy within three weeks of completing the chemotherapy
* Have documented mental disorders
* Have already engaged in other mHealth studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 76 (Actual)
Dates: Start 2022-05-16 (Actual); Primary Completion 2023-08-23 (Actual); Study Completion 2023-08-23 (Actual)

PRIMARY OUTCOMES:
Change from Baseline Score of the Strategies Used by People to Promote Health (SUPPH) at week 3 (T1) and week 6 (T2) | Data collection will be conducted before chemotherapy (baseline), at week 3 (T1), week 6 (T2)
  Strategies Used by People to Promote Health (SUPPH) is a health promotion strategy questionnaire, developed to evaluate the confidence of cancer patients in self-managing their disease, on the basis of expert consultations, patient interviews, and literature research. The original scale has 29 items and uses a 5-point Likert scale, from 1, indicating no confidence to 5, indicating extremely confident. High scores indicate a high level of self-efficacy on the part of the participants. The Chinese version of the SUPPH was adapted by Qian & Yuan and the Cronbach's α coefficient of the total scale is 0.970 . SUPPH will be collected at baseline (week 0), week 3 and at the end of the study (week 6) using self-reported questionnaires handed out through the Breast Health Centre's official WeChat.
Acceptability | Data will be collected at week 6 (T2)
  The intervention acceptability and usability will be tested by a self-report questionnaire, the System Usability Scale, after completing the study (week 6).

SECONDARY OUTCOMES:
Change from Baseline Score of the Functional Assessment of Cancer Therapy-Breast (FACT-B) at week 3 (T1) and week 6 (T2) | Data collection will be conducted before chemotherapy (baseline), at week 3 (T1), week 6 (T2)
  General quality of life has been used as a prominent measurement to reflect the outcome of a treatment. Functional Assessment of Cancer Therapy-Breast (FACT-B) is selected, since it is a HRQoL instrument specific to BC patients. FACT-B is divided into five subscales, namely, physical well-being, social/family well-being, emotional well-being, functional well-being, and additional concerns. Higher scores indicate a better QOL on the part of the participants. Wan et al. reported that the internal consistency of most domains in the simplified Chinese version of FACT-B ranged from 0.82 to 0.85. FACT-B will be collected before chemotherapy (baseline), week 3 and at the end of the study (week 6) using self-reported questionnaires handed out through the Breast Health Centre's official WeChat.
Change from Score at week 3 (T1) of the Memorial Symptom Assessment Scale-Short Form (MSAS-SF) at week 6 (T2) | Data collection will be conducted at week 3 (T1) and week 6 (T2)
  The Memorial Symptom Assessment Scale-Short Form (MSAS-SF) is an instrument that can be used to measure BC patient symptoms of distress. This questionnaire is composed of three dimensions: the Physical Symptom dimension (PHYS), the Psychological Symptom dimension (PSYCH), and a Global Distress Index (GDI). It includes 28 items on distress and frequency in the physical symptom dimension and four items in the psychological symptom dimension during the past week. Higher scores mean more frequency, greater severity and higher distress. The simplified Chinese version of the Memorial Symptom Assessment Scale-Short Form (MSAS-SF-SC) has been found to be reliable, with Cronbach's alpha coefficients for the subscales ranging from 0.782 to 0.874. MSAS-SF will be collected at week 3 and at the end of the study (week 6) using self-reported questionnaires handed out through the Breast Health Centre's official WeChat.
Healthcare service utilization | Data collection will be conducted at week 3 (T1) and week 6 (T2)
  Chemotherapy-induced healthcare utilisation for six weeks will be recorded in the pilot study for analysis. Three types of healthcare utilisation will be collected: patient-initiated hotline calls, unplanned visits to the ambulatory clinic, and unscheduled visits to the emergency department. These records of healthcare service will be obtained from the statistics centre of the study hospital.
End-user engagement by patients and nurses | From baseline up to week 6 (T2)
  Data on an individual's six weeks of usage, including log-in frequency and duration of usage of the whole mChemotherapy program, are tracked in the WeChat statistics module of the background thread. Log-in frequency is recorded as the number of times a participant logged into the app for six weeks. The total duration of usage is recorded as the sum of all times in minutes between logging in and logging out.

CONTACTS AND LOCATIONS:
Overall Officials: Nuo Shi, MPH, Principal Investigator — The Hong Kong Polytechnic University; Arkers KC Wong Dr, PhD, Study Chair — The Hong Kong Polytechnic University; Frances KY Wong Prof, PhD, Study Chair — The Hong Kong Polytechnic University; Xiaobin Lai Dr, PhD, Study Director — Fudan University
Locations (1):
- Ruijin Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No
The pilot study outcomes will only be used to publish, with no personal information revealed. All participant names will be replaced with participant codes to ensure confidentiality and anonymity.

REFERENCES:
- [Background] Bandura A. Self-efficacy: toward a unifying theory of behavioral change. Psychol Rev. 1977 Mar;84(2):191-215. doi: 10.1037//0033-295x.84.2.191. No abstract available. PMID 847061
- [Background] Brady MJ, Cella DF, Mo F, Bonomi AE, Tulsky DS, Lloyd SR, Deasy S, Cobleigh M, Shiomoto G. Reliability and validity of the Functional Assessment of Cancer Therapy-Breast quality-of-life instrument. J Clin Oncol. 1997 Mar;15(3):974-86. doi: 10.1200/JCO.1997.15.3.974. PMID 9060536
- [Background] Chang VT, Hwang SS, Feuerman M, Kasimis BS, Thaler HT. The memorial symptom assessment scale short form (MSAS-SF). Cancer. 2000 Sep 1;89(5):1162-71. doi: 10.1002/1097-0142(20000901)89:53.0.co;2-y. PMID 10964347
- [Background] Fu L, Hu Y, Lu Z, Zhou Y, Zhang X, Chang VT, Yang Y, Wang Y. Validation of the Simplified Chinese Version of the Memorial Symptom Assessment Scale-Short Form Among Cancer Patients. J Pain Symptom Manage. 2018 Jul;56(1):113-121. doi: 10.1016/j.jpainsymman.2018.03.024. Epub 2018 Apr 5. PMID 29627566
- [Background] Lev EL, Owen SV. A measure of self-care self-efficacy. Res Nurs Health. 1996 Oct;19(5):421-9. doi: 10.1002/(SICI)1098-240X(199610)19:53.0.CO;2-S. PMID 8848626
- [Background] Oliveira IS, da Cunha Menezes Costa L, Fagundes FR, Cabral CM. Evaluation of cross-cultural adaptation and measurement properties of breast cancer-specific quality-of-life questionnaires: a systematic review. Qual Life Res. 2015 May;24(5):1179-95. doi: 10.1007/s11136-014-0840-3. Epub 2014 Nov 13. PMID 25391488
- [Background] Yuan C, Qian H, Wang J, Lev EL, Yuan A, Hinds PS. Factorial structure of a scale: Strategies Used by People to Promote Health--Chinese version. Cancer Nurs. 2015 Jan-Feb;38(1):E13-20. doi: 10.1097/NCC.0000000000000151. PMID 24945261
- [Background] Wan C, Zhang D, Yang Z, Tu X, Tang W, Feng C, Wang H, Tang X. Validation of the simplified Chinese version of the FACT-B for measuring quality of life for patients with breast cancer. Breast Cancer Res Treat. 2007 Dec;106(3):413-8. doi: 10.1007/s10549-007-9511-1. Epub 2007 Mar 22. PMID 17377841
- [Derived] Shi N, Ching Wong AK, Yuet Wong FK, Zhang N, Zhu W, Shen K, Lai X, Jin Y, Gu C, Nie L, Dong X. Feasibility of a mobile health app-based self-management program for Chinese patients with breast cancer receiving chemotherapy: A randomized controlled pilot study. Digit Health. 2024 Feb 25;10:20552076241231560. doi: 10.1177/20552076241231560. eCollection 2024 Jan-Dec. PMID 38410790